CLINICAL TRIAL: NCT04712721
Title: Phase I, Open-label, Multicenter Study to Evaluate the Imaging Performance, Safety, Biodistribution and Dosimetry of [68Ga]-FF58 in Adult Patients With Selected Solid Tumors Expected to Overexpress αvβ3 and αvβ5 Integrins.
Brief Title: Study of [68Ga]-FF58 in Patients With Selected Solid Tumors Expected to Overexpress αvβ3 and αvβ5 Integrins.
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CAAA504A12101; 2020-004038-39 (EudraCT Number)
Record Dates: First submitted 2020-12-11; First posted 2021-01-15 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Glioblastoma Multiforme; Brain Neoplasms; Gastroesophageal Adenocarcinoma; Pancreatic Ductal Adenocarcinoma
Keywords: Glioblastoma Multiforme; GBM; Breast Cancer; BC; Brain Metastasis from BC; Gastroesophageal adenocarcinoma; GEA; Pancreatic ductal adenocarcinoma; PDAC; alpha-v beta 3 integrin; αvβ3; alpha-v beta 5 integrin; αvβ5; Dosimetry; 68Gallium; 68Ga; FF58; [68Ga]-FF58
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Imaging study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Glioblastoma Multiforme (Experimental): All eligible participants will receive recommended dose of [68Ga]-FF58 of 3 Megabecquerel (MBq)/Kg (+/- 10%) [but not more than 250 and not less than 150 MBq].
  Interventions: Drug: 68Ga-FF58
- Brain Metastasis from Breast Cancer (Experimental): All eligible participants will receive recommended dose of [68Ga]-FF58 of 3 Megabecquerel (MBq)/Kg (+/- 10%) [but not more than 250 and not less than 150 MBq].
  Interventions: Drug: 68Ga-FF58
- Gastroesophageal adenocarcinoma (Experimental): All eligible participants will receive recommended dose of [68Ga]FF58 of 3 Megabecquerel (MBq)/Kg (+/-10%) [but not more than 250 and not less than 150 MBq]
  Interventions: Drug: 68Ga-FF58
- Pancreatic ductal adenocarcinoma (Experimental): All eligible participants will receive recommended dose of [68Ga]FF58 of 3 Megabecquerel (MBq)/Kg (+/-10%) [but not more than 250 and not less than 150 MBq]
  Interventions: Drug: 68Ga-FF58

INTERVENTIONS:
Drug: 68Ga-FF58 — Single intravenous radiolabeled gallium FF58 injection determined by body weight (3 Megabecquerel (MBq)/Kg (+/- 10%)). Administered dose must not be lower than 150 MBq or higher than 250 MBq.

SUMMARY:
This is a First-In-Human (FIH) study of [68Ga]-FF58 to characterize the imaging properties, safety, biodistribution and dosimetry properties of [68Ga]-FF58 in adults with relapsed or refractory (r/r) glioblastoma multiforme (GBM), breast cancer (BC) that has metastasized to the brain, gastroesophageal adenocarcinoma (GEA) or pancreatic ductal adenocarcinoma (PDAC) expected to overexpress alpha-v beta 3 (αvβ3) and alpha-v beta 5 (αvβ5) integrins.

DETAILED DESCRIPTION:
Approximately 80 patients were planned to be enrolled into the study, 20 patients with GBM, 20 patients with BC that had metastasized to the brain, 20 with GEA and 20 with PDAC.

The study included an imaging characterization part and an expansion part. In the imaging characterization part, approximately 24 patients were planned to be enrolled, 6 with r/r GBM, 6 with BC that had metastasized to the brain, 6 with GEA and 6 with PDAC. Due to the early termination of the study, the expansion part was not started.

Both parts of the study (imaging characterization and expansion) included a dosimetry sub-group in which the distribution, pharmacokinetics (PK), radiation dosimetry and absorbed doses in tissue and tumor were to be assessed. However, no patients were enrolled in the dosimetry sub-group.

All patients enrolled in the study received a single dose of [68Ga]-FF58 and underwent [68Ga]-FF58 positron emission tomography (PET) imaging at different timepoints on Day 1 as well as conventional imaging (high resolution computed tomography (CT) or magnetic resonance imaging (MRI)).

The estimated study duration for each individual patient was approximately 44 days (including screening period of 28 days and 14 days of follow-up (FU)).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study
* Patients with histologically or cytologically confirmed and documented r/r GBM that has progressed after prior radiation therapy and have not received prior bevacizumab OR patients with BC that has metastasized to the brain and who should have at least one newly diagnosed brain metastasis that has not been resected or irradiated, or has been irradiated and progressed OR patients with histologically or cytologically confirmed and documented locally advanced or metastatic GEA (i.e., adenocarcinoma of the stomach (intestinal subtype), esophagus, or gastroesophageal junction), either untreated or r/r after one or more lines of treatment OR patients with histologically or cytologically confirmed and documented locally advanced or metastatic PDAC, either untreated or r/r after one or more lines of treatment.

Exclusion Criteria:

* Creatinine clearance (calculated using Cockcroft-Gault formula) <40 mL/min.
* Unmanageable bladder outflow obstruction or urinary incontinence.
* QTcF > 480 msec on screening ECG or congenital long QT syndrome.
* Any condition that requires chronic treatment with anticoagulants or antiplatelet agents
* Patients with a known bleeding disorder
* Administration of a radiopharmaceutical within a period corresponding to 10 half-lives of the radionuclide used prior to injection of [68Ga]-FF58.
* Pregnant women. Women who are breastfeeding must express and discard breast milk for 12 hours after [68Ga]-FF58 administration and must also stop breast feeding during this same period. Males and females must abstain from sexual intercourse for 12 hours after [68Ga]-FF58 administration.
* Total bilirubin > 1.5 x ULN (except for patients with Gilbert's syndrome who are excluded if total bilirubin > 3.0 x ULN) or direct bilirubin > 1.5 x ULN
* Alanine aminotransferase (ALT) > 3 x ULN, except for patients that have tumor involvement of the liver, who are excluded if ALT > 5 x ULN
* Aspartate aminotransferase (AST) > 3 x ULN, except for patients that have tumor involvement of the liver, who are excluded if AST > 5 x ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Time-activity curves (TACs) from 68Ga-FF58 PET/CT images | [68Ga]-FF58 PET imaging acquired at Day 1
  Time activity curves (TACs) for the various organs will be produced as mean Standard Uptake Values (SUV) of the lesions over time.
Standard Uptake Value (SUV) mean and max in lesions detected by PET scans | [68Ga]-FF58 PET imaging acquired at Day 1
  Targeting properties of 68GaFF58 will be evaluated by semi quantitatively assessing radiotracer uptake at lesion level, identified via PET/CT imaging (4 scans). The SUVmean and SUVmax of each lesion will be calculated and reported by lesion location with summary statistics.
Tumor to Background Ratio (TBR) of lesions detected by PET scans | [68Ga]-FF58 PET imaging acquired at Day 1
  Targeting properties of 68Ga-FF58 will be evaluated by semi quantitatively assessing radiotracer uptake at lesion level, identified via PET/CT imaging (4 scans). The lesion Tumor to Background Ratio (TBR) will be defined as the ratio of the lesion SUV over the reference region SUV. TBRs will be calculated for both SUVmax(lesion) / SUVmean and reported by lesion location with summary statistics. Different regions will be used as reference, in order to satisfy the most appropriate one for each type of lesion.

SECONDARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events | From first dosing (single administration, Day 1) up to 14 days post infusion
  Treatment-emergent adverse events (TEAEs) will be collected from first dosing (single administration, Day 1) up to last follow-up visit or the patient withdrew consent. The distribution of adverse events will be done via the analysis of frequencies for treatment emergent Adverse Event (TEAEs), Serious Adverse Event (TESAEs) and Deaths due to AEs, through the monitoring of relevant clinical and laboratory safety parameters.
Percentage of lesions detected by conventional scans, PET scans, or both modalities | [68Ga]-FF58 PET imaging acquired at Day 1
  The percentage of lesions detected by conventional imaging (high resolution CT or MRI acquired jointly or within 24 hours before or after the [68Ga]-FF58 PET scan), [68Ga]-FF58 PET scans , or both modalities will be summarized descriptively for all patients and split by indication.
Lesion-level analyses of diagnostics by [68Ga]-FF58 compared with conventional imaging | [68Ga]-FF58 PET imaging acquired at Day 1
  At lesion level, overall, positive, and negative agreement of [68Ga]-FF58 will be calculated based on the aforementioned tabulations as follows: • Overall agreement = 100% x (Double positive + Double negative) / total number of lesions identified by either imaging procedures
  * Positive agreement = 100% x Double positive / (Double positive + Comparator single positive)
  * Negative agreement = 100% x Double negative / (Double negative + Comparator single negative).
Dosimetry Group: Area under the serum concentration-time curve from time zero to the time of last quantifiable concentration (AUClast) of 68Ga-FF58 | Day 1 (0, 0-5, 10, 30, 60, 120, 180-240, 300 minutes post infusion)
  Venous whole blood samples will be collected and analysed for radioactivity. Radioactivity-based concentration units will be converted to mass-based concentration units using the specific activity of the dose at the time of manufacture (MBq/µg). Pharmacokinetics characterization will be performed on mass-based concentrations. AUClast will be listed and summarized using descriptive statistics.
Dosimetry Group: Time of maximum observed drug concentration occurrence (Tmax) of 68Ga-FF58 | Day 1 (0, 0-5, 10, 30, 60, 120, 180-240, 300 minutes post infusion)
  Venous whole blood samples will be collected and analysed for radioactivity. Radioactivity based concentration units will be converted to mass-based concentration units using the specific activity of the dose at the time of manufacture (MBq/µg). Pharmacokinetics characterization will be performed on mass-based concentrations. Tmax will be listed and summarized using descriptive statistics.
Dosimetry Group: Observed maximum plasma concentration (Cmax) of 68Ga-FF58 | Day 1 (0, 0-5, 10, 30, 60, 120, 180-240, 300 minutes post infusion)
  Venous whole blood samples will be collected and analysed for radioactivity. Radioactivity based concentration units will be converted to mass-based concentration units using the specific activity of the dose at the time of manufacture (MBq/µg). Pharmacokinetics characterization will be performed on mass-based concentrations. Cmax will be listed and summarized using descriptive statistics.
Dosimetry Group: Terminal elimination half-life (T^1/2) of 68Ga-FF58 | Day 1 (0, 0-5, 10, 30, 60, 120, 180-240, 300 minutes post infusion)
  Venous whole blood samples will be collected and analysed for radioactivity. Radioactivity based concentration units will be converted to mass-based concentration units using the specific activity of the dose at the time of manufacture (MBq/µg). Pharmacokinetics characterization will be performed on mass-based concentrations. The half-life will be listed and summarized using descriptive statistics.
Dosimetry Group: Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUCinf) of 68Ga-FF58 | Day 1 (0, 0-5, 10, 30, 60, 120, 180-240, 300 minutes post infusion)
  Venous whole blood samples will be collected and analysed for radioactivity. Radioactivity based concentration units will be converted to mass-based concentration units using the specific activity of the dose at the time of manufacture (MBq/µg). Pharmacokinetics characterization will be performed on mass-based concentrations. AUCinf will be listed and summarized using descriptive statistics.
Dosimetry Group: Total systemic clearance for intravenous administration (CL) of 68Ga-FF58 | Day 1 (0, 0-5, 10, 30, 60, 120, 180-240, 300 minutes post infusion)
  Venous whole blood samples will be collected and analysed for radioactivity. Radioactivity based concentration units will be converted to mass-based concentration units using the specific activity of the dose at the time of manufacture (MBq/µg). Pharmacokinetics characterization will be performed on mass-based concentrations. CL will be listed and summarized using descriptive statistics.
Dosimetry Group: Volume of distribution during the terminal phase following intravenous elimination (Vz) of 68Ga-FF58 | Day 1 (0, 0-5, 10, 30, 60, 120, 180-240, 300 minutes post infusion)
  Venous whole blood samples will be collected and analysed for radioactivity. Radioactivity based concentration units will be converted to mass-based concentration units using the specific activity of the dose at the time of manufacture (MBq/µg). Pharmacokinetics characterization will be performed on mass-based concentrations. Vz will be listed and summarized using descriptive statistics.
Dosimetry Group: Urinary excretion of radioactivity expressed as a percentage of injected activity (%IA) | Day 1 (0-30, 30-120, 120-180, 180-300 minutes post infusion)
  Urine samples will be collected over specified time intervals and analysed for radioactivity. The radioactivity excreted in each interval as a percentage of injected activity (%IA) will be listed and summarized using descriptive statistics.
Dosimetry Group: Absorbed dose of 68Ga- FF58 | [68Ga]-FF58 PET imaging acquired at Day 1
  The absorbed dose in target organs will be summarized with descriptive statistics. Lesion number will be assigned by dosimetry expert.
Dosimetry Group: Effective whole-body dose of 68Ga- FF58 | [68Ga]-FF58 PET imaging acquired at Day 1
  The effective radiation dose will be summarized with descriptive statistics. Lesion number will be assigned by dosimetry expert.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Investigative Site, Lyon, France
- Novartis Investigative Site, Essen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18293
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2579